CLINICAL TRIAL: NCT05456594
Title: Comparing Sports Bra Design in Full Busted Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: Bounceless (Unknown)
Responsible Party: Principal Investigator, Stacey Gorniak, Associate Professor, University of Houston
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00003644
Record Dates: First submitted 2022-06-29; First posted 2022-07-13 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Breast Pain; Mastalgia; Back Pain; Back Strain; Back Pain, Low; Neck Pain; Chest Pain; Activity, Motor; Aging Well; Weight, Body; Body Image
MeSH Terms: conditions — Mastodynia; Back Pain; Low Back Pain; Neck Pain; Chest Pain; Motor Activity; Body Weight

STUDY DESIGN:
Intervention Model Description: This study involves use of a cross-sectional observation and analysis of behavior using a cross-over approach in assessing 2 sports bra models.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional bra (Placebo Comparator): Measurement of kinematic and kinetic data during physical activities while participant is wearing their own conventional bra.
  Interventions: Other: Bounceless bra; Other: Shefit bra
- Bounceless bra (Active Comparator): Measurement of kinematic and kinetic data during physical activities while participant is wearing provided Bounceless bra.
  Interventions: Other: Conventional bra; Other: Shefit bra
- Shefit bra (Active Comparator): Measurement of kinematic and kinetic data during physical activities while participant is wearing provided Shefit bra.
  Interventions: Other: Conventional bra; Other: Bounceless bra

INTERVENTIONS:
Other: Conventional bra — This study involves use of a cross-sectional observation and analysis of behavior using a cross-over approach in assessing breast motion while using a conventional bra (bra condition #1).
  Arms: Bounceless bra; Shefit bra
Other: Bounceless bra — This study involves use of a cross-sectional observation and analysis of behavior using a cross-over approach in assessing breast motion while using a provided Bounceless bra (bra condition #2a).
  Arms: Conventional bra; Shefit bra
Other: Shefit bra — This study involves use of a cross-sectional observation and analysis of behavior using a cross-over approach in assessing breast motion while using a provided Shefit bra (bra condition #2b).
  Arms: Bounceless bra; Conventional bra

SUMMARY:
The goal of the current project is to assess performance of the Bounceless Control sports bra versus: (1) the Shefit Ultimate Sports bra, and (2) conventional bra as worn by participants in a variety of athletic activities.

DETAILED DESCRIPTION:
Research has shown that during activities such as running and jumping, bare breasts move up and down as much as 12 cm. This is due to insufficient anatomical support within the breasts (https://sma.org.au/resources-advice/injury-fact-sheets/exercise-and-breast-support/).

Conventional bras do not provide enough breast support during athletic activities. Additionally, dynamic breast movement induces motion/slippage of conventional bra straps, skin chaffing due to friction, and skin irritation/abrasion/soreness due to impression of metal fixtures (e.g., hooks, underwires, etc.) within the bras. In response to the inadequacies of conventional bras, the first sports bras were invented in 1977. The sports bra (originally known as the "Jogbra") is considered a groundbreaking item which helped remove a major barrier to women's participation in athletic activities. The original Jogbra was created by sewing 2 mens athletic supports together.

While the design of Jogbra was simple in its original form, updates to modern materials and sewing techniques over the past 45 years has spawned a wide variety of sports bras that are available worldwide. Modern sports bras vary in materials and construction techniques. These features dictate the sizes available for the bras was well as recommended uses for the bras. Most commercially available sport bras are designed for low to medium impact activities in sizes ranging from extra small (US bra size 32A) to extra large (40C). The design of most of these sports bras are similar to the original Jogbra design.

Despite the availability of sports bras in many sizes, materials, and constructions, women with larger breasts (cup sizes C+) still experience excessive breast movement during exercise, even while wearing a sports bra. Such movement is uncomfortable and may be embarrassing. Both breast discomfort and embarrassment are recognized as significant barriers to physical activity in women. Women with larger breast sizes thus require greater support from their sports bra (https://sma.org.au/resources-advice/injury-fact-sheets/exercise-and-breast-support/).

Unfortunately, due to the commercial desire to keep costs as low as possible in production of sports bras, the materials and designs used in most sports bras remain inadequate for women with larger breast sizes. In many cases, women with larger breast continue to wear a conventional bra underneath a sports bra or 2 sports bras together for increased breast support during athletic activities.

Recently, 2 companies (Shefit and Bounceless) have attempted to address this issue in the marketplace. Shefit is the larger of the 2 companies working to offer more supportive sports bra options. A recent study of sports bra performance in women with breast sizes ranging from AA-DD found that the Shefit Ultimate Sports bra performed similar to other sports bras offered by large manufacturers of athletic equipment (e.g., Nike, Underarmor) (Gibson et al. 2019). The Bounceless project was omitted from such testing. The Bounceless Control sports bra offers additional support beyond the Shefit Ultimate Sports bra as it is a long line (additional fabric that extends below the bust) sports bra with an internal breast band to support breasts during activity while also preventing multidirectional accelerations of breast material during activity.

The goal of the current project is to assess performance of the Bounceless Control sports bra versus: (1) the Shefit Ultimate Sports bra, and (2) conventional bra as worn by participants in a variety of athletic activities.

References:

Gibson TM, Balendra N, Ustinova KI, Langenderfer JE. Reductions in Kinematics from Brassieres with Varying Breast Support. International Journal of Exercise Science. 2019;12(1):402-411.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Age of 18 to 55 years
3. Female sex at birth
4. Self-declared breast size of D-G cup (US sizes: D, DD/E, DDD/F, DDDD/G)
5. Bra band size between 32-40"
6. International Physical Activity Questionnaire - Short Form (IPAQ-SF) score of 3 or higher
7. An answer of "NO" to any item of the general health questions of the PARQ+
8. No history of surgery to: back, neck, or shoulders
9. No history of breast reconstruction
10. No history of spinal cord injury (SCI)

Exclusion Criteria:

1. Inability to provide informed consent
2. Age 17 years old or younger or 56 years or older
3. Male sex at birth

k. Self-declared breast size of smaller than D cup or larger than G cup (US sizes) d. Bra band size outside of the range 32-40" e. IPAQ-SF score of 2 or lower f. An answer of "YES" to any item of the general health questions of the PARQ+ g. Diagnosis of Type I Diabetes, Diagnosis of Type II Diabetes, Type III Diabetes, Latent Autoimunne diabetes in adults (LADA), or current Gestational Diabetes h. History of limb amputation (upper or lower extremity) i. Presence of open pressure sores on the upper or lower extremities j. History of breast augmentation, reconstruction, or mastectomy k. Currently pregnant or lactating/breastfeeding l. History of surgery to: back, neck, or shoulders m. History of the following neurological diseases: Cerebrovascular accident (CVA, stroke), Alzheimer's Disease (AD), Dementia (of any form), Huntington's Disease, Traumatic Brain Injury (TBI), Spinal cord injury (SCI), Multiple Sclerosis (MS), Parkinson's Disease (PD), Polio, Paraproteinaemic Demyelinating Neuropathy (PDN) and/or Monoclonal Gammopathy of Undetermined Significance (MGUS), Myasthenia Gravis, Muscular Dystrophy, Rheumatoid Arthritis, Guillain-Barré Syndrome, Charcot-Marie-Tooth Disorder or other hereditary neuropathies, or pain in the extremities (shoulder, elbows, wrist, fingers, hips, knees, ankles, or feet) that severely limit activities of daily living.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Biomechanical Data | 1 day
  Segmental displacement (m)
Biomechanical Data | 1 day
  Segmental velocity (m/s)
Biomechanical Data | 1 day
  Segmental acceleration (m/s^2)
Biomechanical Data | 1 day
  Gait speed (m/s)
Biomechanical Data | 1 day
  Cadence (Hz)
Biomechanical Data | 1 day
  Muscle activity (mV)
Pain Measures | 1 day
  Qualitative assessment of pain via self report (no units)

SECONDARY OUTCOMES:
Anthropometry | 1 day
  Height (m)
Anthropometry | 1 day
  Mass (kg)
Anthropometry | 1 day
  Percent body fat (%)
Glycated Hemoglobin | 1 day
  A1c (%)
Sex-Hormones | 1 day
  Estrone (mg/dL)
Sex-Hormones | 1 day
  Estradiol (mg/dL)
Sex-Hormones | 1 day
  Testosterone (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Online Screening Form for Potential Participants — https://universityofhouston.iad1.qualtrics.com/jfe/form/SV_9M6NXHOFjYLm38G